CLINICAL TRIAL: NCT06109948
Title: A Phase 1a/1b, Single Ascending Dose and Multiple Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ABX1100 in Normal Healthy Volunteers and Late-onset Pompe Disease Patients
Brief Title: Study to Assess the Safety, Tolerability, PK and PD of ABX1100
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Aro Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABX1100-1001
Record Dates: First submitted 2023-10-19; First posted 2023-10-31 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Healthy; Late Onset Pompe Disease
Keywords: pompe; GYS1
MeSH Terms: interventions — Infusions, Intravenous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A Cohort 1-4 Single Dose (active) (Experimental): Subjects will receive 1 single IV dose of ABX1100 on Day 1.
  Interventions: Drug: ABX1100 injection for IV infusion
- Part A Cohort 1-3 Single Dose (placebo) (Placebo Comparator): Subjects will receive 1 single IV dose of placebo on Day 1.
  Interventions: Drug: Placebo injection for IV infusion
- Part B Multi-dose (active) (Experimental): Subjects will receive 1 IV dose of ABX1100 on Day 1 and Day 29 each.
  Interventions: Drug: ABX1100 injection for IV infusion
- Part B Multi-dose (placebo) (Placebo Comparator): Subjects will receive 1 IV dose of placebo on Day 1 and Day 29 each.
  Interventions: Drug: Placebo injection for IV infusion
- Part C (Experimental): Late onset Pompe Disease patients will receive 1 dose of ABX1100 at Day 1 and Day 29 respectively.
  Interventions: Drug: ABX1100 injection for IV infusion

INTERVENTIONS:
Drug: ABX1100 injection for IV infusion — Centyrin protein-siRNA conjugate
  Arms: Part A Cohort 1-4 Single Dose (active); Part B Multi-dose (active); Part C
Drug: Placebo injection for IV infusion — placebo saline injection
  Arms: Part A Cohort 1-3 Single Dose (placebo); Part B Multi-dose (placebo)

SUMMARY:
Study ABX1100-1001 is a first-in-human (FIH), phase 1 study to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of a single ascending dose (SAD) and multiple doses (MD) of ABX1100 administered intravenously to healthy participants and patients with LOPD.

* Part A features a SAD study with a double-blind, placebo-controlled, randomized design in NHVs involving 3 cohorts (A1-A3). This Part also includes a single dose, open-labeled cohort (A4) in NHVs which will commence after cohorts A1-3.
* Part B is a MD, double-blind, placebo-controlled, randomized design in NHVs. The MD Part B will commence after completion of Cohorts A1, A2 and A3 in the SAD Part A and SRC review of these 3 cohorts.
* Part C opened for enrollment after the Safety Review Committee (SRC) review of safety, PK and PD data from both Part A and Part B. Part C is a MD, open-label design in patients with Late-Onset Pompe Disease.

ELIGIBILITY:
Parts A-B Inclusion Criteria:

* Body mass index (BMI) between 18.0 and 32.0 kg/m2, inclusive and weight between 50 and 90 kg, inclusive.
* Agree not to have a tattoo or body piercing until the end of the study.
* Agree not to receive COVID-19 vaccination from 7 days prior to first study drug administration until at least 7 days after the last study drug administration.
* Agree not to receive a vaccination (live attenuated vaccine) during the study and until 60 days after the study has ended (last study procedure).
* Willing to undergo needle muscle biopsies.
* Willing to avoid strenuous activities 48 hours before needle muscle biopsy and throughout the study.
* Female participants who are sexually active with a non-sterilized partner must be non-pregnant and non-lactating and agree to use a highly effective method of contraception.
* Males of childbearing potential must agree to use a highly effective method of contraception with female sexual partners of childbearing potential and not donate sperm during study participation and for 90 days after last administration of study drug ABX1100 or placebo.

Parts A-B Exclusion Criteria:

* Known history or presence of any clinically significant hepatic, renal/genitourinary, gastrointestinal, cardiovascular, cerebrovascular, pulmonary, endocrine, immunological, musculoskeletal, neurological, psychiatric, dermatological or hematological disease or condition.
* History of any inherited or acquired skeletal muscle diseases (for example, Duchenne Muscular Dystrophy (DMD), Becker Muscular Dystrophy (BMD), Limb-Girdle Muscular Dystrophy (LGMD), Myotonic Dystrophy, Spinal Muscular Atrophy (SMA), Polymyositis, Rhabdomyolysis and Inclusion Body Myositis (IBM).
* History of any inherited or acquired cardiac disease including congestive heart failure, ischemic heart disease, or arrhythmias; an abnormal ECG.
* History of cancer within past 5 years, with the exception of treated or excised skin basal cell carcinoma.
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks prior to the screening visit
* Presence of any significant physical or organ abnormality.
* Major surgery within 6 months prior to the start of the study.
* Current smoker, recent history of smoking and/or use of any nicotine-containing products (within past 6 months).
* A known history or positive test result for hepatitis B surface antigen (HBsAg), hepatitis C antibody or human immunodeficiency virus (HIV) infection.
* Currently participating in another investigational trial or have received any investigational drug within the past 30 days.

Part C Key Inclusion criteria

* Male or female LOPD patients aged ≥ 18 years (inclusive) of age, at the time of informed consent.
* Body mass index (BMI) between 18.0 and 35.0 kg/m2, inclusive and weight >50 kg.
* Agree not to receive COVID-19 vaccination from 7 days prior to first study drug administration until at least 7 days after the last study drug administration or after the final study procedure, whichever is later.
* Agree not to receive a vaccination (live attenuated vaccine) during the study and until 60 days after the study has ended (last study procedure).
* Willing to undergo needle muscle biopsies.
* Documented Acid alpha-glucosidase (GAA) deficiency and mutation analysis from blood, skin, or muscle tissue for confirmation of diagnosis of LOPD.
* Currently receiving a stable dose of standard of care enzyme replacement therapy (ERT) regularly for a minimum of 6 months immediately prior to study entry
* Capable of walking 50 meters with or without an assistive device.
* Predicted upright Forced Vital Capacity (FVC) >= 30% within the past year prior to study entry, not requiring invasive mechanical ventilation. Non-invasive, temporary, respiratory support is acceptable
* Female participants who are sexually active with a non-sterilized partner must be non-pregnant and non-lactating and agree to use a highly effective method of contraception.
* Males of childbearing potential must agree to use a highly effective method of contraception with female sexual partners of childbearing potential and not donate sperm during study participation and for 90 days after last administration of study drug ABX1100.

Part C Key Exclusion criteria

* History of muscle biopsy within 1 month of Day 1 or planning to undergo non-study related muscle biopsies during study period.
* History of coronary artery disease or cardiovascular disease.
* History or presence of gastrointestinal, renal, or hepatic disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Presence of any significant physical or organ abnormality as determined by the PI/Sub-Investigator.
* Resting seated blood pressure < 90/40 mmHg or > 140/90 mmHg , unless deemed not clinically significant by the PI/Sub-Investigator.
* Resting seated heart rate < 45 bpm or > 99 bpm, unless deemed not clinically significant by the PI/Sub-Investigator.
* Intolerance to and/or difficulty with blood sampling through venipuncture.
* Positive pregnancy test for female participants.
* Currently participating in another investigational trial or have received any investigational drug within the past 30 days or 5 elimination half-lives of the investigational drug, whichever is longer, prior to dosing.
* Requires a wheelchair or invasive ventilation.
* Fridericia's corrected QT (QTcF) > 450 ms for participants or history of QT interval prolongation unless deemed not clinically significant by the PI/Sub-Investigator.
* Uncontrolled diabetes (Hemoglobin A1c [HbA1c] equal to or higher than 7.5%).
* A known history or positive test result for hepatitis B surface antigen (HBsAg), hepatitis C antibody or human immunodeficiency virus (HIV) infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-10-19 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with treatment-emergent adverse events (TEAEs) | up to 20 weeks
  Adverse Events will be graded in accordance with the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 5.0. Adverse events (AEs) will be reported based on clinical laboratory tests, vital signs, physical examinations, electrocardiograms, and echocardiograms from the time informed consent is signed through 8 weeks after ABX1100 administration for Part A and through 12 weeks after ABX1100 administration for Part B, and up to 20 weeks for Part C. AEs will be considered to be treatment emergent (TEAE) if they occurred or worsened in severity after the first dose of study treatment.

SECONDARY OUTCOMES:
Plasma pharmacokinetics as measured by Cmax | 0-8 hours after ABX1100 administration
  Plasma samples will be taken pre-dose, 10 min, end of infusion, 0.5, 1, 3, 6 and 8 hours after the start of ABX1100 administration
Plasma pharmacokinetics as measured by Tmax | 0-8 hours after ABX1100 administration
  Plasma samples will be taken pre-dose, 10 min, end of infusion, 0.5, 1, 3, 6 and 8 hours after the start of ABX1100 administration
Plasma pharmacokinetics as measured by AUC | 0-8 hours after ABX1100 administration
  Plasma samples will be taken pre-dose, 10 min, end of infusion, 0.5, 1, 3, 6 and 8 hours after the start of ABX1100 administration
Immunogenicity of AXB1100 as measured by anti-ABX1100 antibodies in serum | Up to 16 weeks
  Plasma samples will be taken pre-dose, Day 15 and Day 29 after ABX1100 administration (Part A); Plasma samples will be taken pre-dose, Day 15, Day 29, Day 43, Day 57 and Day 71 after ABX1100 administration (Part B); Plasma samples will be taken pre-dose, Day 15, Day 29, Day 43, Day 57 and Day 71 after ABX1100 administration; D113 blood draw for ADA may be requested by Sponsor based on results of earlier timepoints. (Part C);
Muscle drug concentration | Needle muscle biopsies at pre-dose, week 10 and week 6 or 16
  Concentration of siRNA component in skeletal muscle
Pharmacodynamics as measured by GYS1 mRNA in muscle | Needle muscle biopsies at pre-dose, week 10 and week 6 or 16
  Change in GYS1 mRNA from pre-dose

CONTACTS AND LOCATIONS:
Locations (5):
- United States (3):
  - UCI, Orange, California
  - Washington University School of Medicine, St Louis, Missouri
  - Lysosomal and Rare Disorders Research and Treatment Center, Inc, Fairfax, Virginia
- Canada (2):
  - MAGIC clinic, Calgary, Alberta
  - McMaster University, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No